CLINICAL TRIAL: NCT01694953
Title: The Rare Disease Clinical Research Network Natural History Study of MNGIE
Brief Title: The Natural History Study of Mitochondrial NeuroGastroIntestinal Encephalopathy (MNGIE)
Acronym: NAHIM
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAI5453; 1U54NS078059 (NIH)
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Mitochondrial NeuroGastroIntestinal Encephalopathy (MNGIE)
Keywords: MNGIE; Mitochondrial; Mitochondrial Neurogastrointestinal encephalopathy
MeSH Terms: conditions — Visceral myopathy familial external ophthalmoplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with MNGIE: Patients of all races of any gender who are at least 5 years of age with a defect in thymidine phosphorylase may participate in this natural history study.

SUMMARY:
This is a multi-center natural history study of Mitochondrial NeurogastroIntestinal Encephalopathy (MNGIE). Patients will be followed over time to assess clinical symptoms. The investigators hope to learn more about the disease of MNGIE as well as develop useful measures of disease status for use in future clinical trials.

Additional clinical centers will be listed as they become available.

DETAILED DESCRIPTION:
The investigators will examine a total of 20 patients at six month intervals for up to five years. The investigators will evaluate gastrointestinal function, lean body mass, neuropathy, neuropsychological capability, quality of life, nutrition, motor function and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Thymidine Phosphorylase (TP) defect:

   1. homozygous or
   2. compound heterozygous mutations in the TYMP gene, and/or
   3. TP enzyme activity of <20% of normal.
2. Increased plasma Thd > 3 micromole/L
3. Increased plasma dUrd > 7.5 micromole/L
4. Age requirement of at least 5 years of age.

Exclusion Criteria:

1. Participation in an interventional (study medication or other experimental intervention) study (within 1 month of participation in this study).
2. Unable to travel to site for research visits.
3. Unwillingness to sign informed consent form.
4. Substance abuser

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female, At least 5 years of age, with Thymidine Phosphorylase defect
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Timed Water Swallow | 5 years
  The timed water swallow test evaluates the time it takes to swallow a small cup of water

SECONDARY OUTCOMES:
Degree of Neuropathy | 5 years
  A general neurological exam will be performed to assess the degree of neuropathy.

OTHER OUTCOMES:
Score on Mini Mental State Exam | 5 years
  A short assessment of cognitive function will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
When applicable manuscript(s) will be submitted.
Time Frame: When applicable manuscript(s) will be submitted.
Access Criteria: Data included in manuscript(s).

REFERENCES:
- [Background] Marti R, Lopez LC, Hirano M. Assessment of thymidine phosphorylase function: measurement of plasma thymidine (and deoxyuridine) and thymidine phosphorylase activity. Methods Mol Biol. 2012;837:121-33. doi: 10.1007/978-1-61779-504-6_8. PMID 22215544
- See also: Rare Disease Clinical Research Network, NIH — https://www.rarediseasesnetwork.org/